CLINICAL TRIAL: NCT05468528
Title: Clinical Value of Linear Ablation Without Pulmonary Vein Isolation in Persistent Atrial
Brief Title: Clinical Value of Linear Ablation Without Pulmonary Vein Isolation in Persistent Atrial Fibrillation
Acronym: CLEAR AF II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); ZHONGNANSHAN MEDICAL FOUNDATION OF GUANGDONG PROVINCE (Unknown); Beijing Hospital (Other Government); Wuhan Asia Heart Hospital (Other); Tianjin Medical University General Hospital (Other); Fuwai Yunnan Cardiovascular Hospital (Other); RenJi Hospital (Other); Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-1627
Record Dates: First submitted 2022-06-14; First posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Atrial Fibrillation, Persistent; Atrial Fibrillation
Keywords: linear ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- linear ablation group (Experimental): The linear ablation is performed on the basis of Ω-type linear ablation. Further stepwise ablation of the left atrial anterior wall increases the blockage of the LA roof and the MVA isthmus. Ablation in CS or ethanol ablation of vein of Marshall. Also, epicardial ablation on the roof or rigid between LAA-LPVs may be applied if necessary.
  Interventions: Procedure: catheter radiofrequency ablation(individualized stepwise linear without pulmonary vein isolation)
- PVI group (Other): pulmonary vein isolation ablation alone
  Interventions: Procedure: catheter radiofrequency ablation(PVI)

INTERVENTIONS:
Procedure: catheter radiofrequency ablation(individualized stepwise linear without pulmonary vein isolation) — individualized stepwise linear ablation without pulmonary vein isolation
  Arms: linear ablation group
Procedure: catheter radiofrequency ablation(PVI) — pulmonary vein isolation
  Arms: PVI group

SUMMARY:
Based on previous theoretical foundation and clinical practice experience, the investigators further propose a multi-center randomized prospective trial to compare the pure linear ablation strategy without pulmonary vein isolation to traditional PVI ablation for persistent AF. population size is 207. The participants will be randomized to the linear ablation group and PVI ablation group with a 2:1 ratio. the follow-up period is 12 months. The primary outcome is freedom from atrial fibrillation, the secondary outcome is complications related to ablation.

DETAILED DESCRIPTION:
Pulmonary vein isolation is recommended as the cornerstone of catheter ablation of atrial fibrillation by current guidelines, However, meta-analysis suggests that the success rate of continuous pulmonary vein isolation for persistent atrial fibrillation is only 43%. Therefore, in addition to pulmonary vein isolation, further research on substrate modification in the treatment of atrial fibrillation is particularly important.

Based on our previous theoretical foundation and clinical practice experience, the investigators further propose a multi-center randomized prospective trial to compare the pure linear ablation strategy without pulmonary vein isolation to traditional PVI ablation for persistent AF. The linear ablation is performed on the basis of Ω-type linear ablation. Further stepwise ablation of the left atrial anterior wall increases the blockage of the LA roof and the MVA isthmus. Ablation in CS or ethanol ablation of vein of Marshall. Also, epicardial ablation on the roof or rigid between LAA-LPVs may be applied if necessary.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from persistent atrial fibrillation and referred to catheter ablation therapy.
* patients agreeing to be enrolled， with the informed consent signed

Exclusion Criteria:

1. Sinus rhythm at the time of recruitment;
2. Age less than 18 years old or older than 75 years;
3. Transthoracic echocardiography suggests that the anteroposterior diameter of the left atrium is greater than 55 mm;
4. History of previous radiofrequency ablation of atrial fibrillation or surgical ablation History;
5. Left atrial thrombus recorded by ultrasound or CT;
6. Combined with severe lung disease;
7. Previous history of cardiac surgery;
8. Patients with hyperthyroidism, atrial septal defect, mitral stenosis, or severe coronary heart disease requiring further treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Freedom from atrial fibrillation at 1 year | 12 months after the ablation
  Recurrent AF is defined as documented AF (through 12-lead ECG) episode lasting >30 seconds after a 3-month blanking period.

SECONDARY OUTCOMES:
complications related to ablation | 12 months after the ablation
  Tamponade, pericarditis and perforation following the ablation procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided